CLINICAL TRIAL: NCT06574204
Title: The Mechanism and Clinical Observations of Pain and Pruritus Induced by Exposure to Allergic Contact Dermatitis Resulting From Macrolides
Brief Title: Clinical Observations of Pain and Pruritus Induced by Exposure to Allergic Contact Dermatitis Caused by Macrolides
Status: Not yet recruiting | Type: Observational
Sponsor: Affiliated Hospital of Nantong University (Other)
Responsible Party: Sponsor
Other Study IDs: LCYJ20242026
Record Dates: First submitted 2024-08-25; First posted 2024-08-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Dermatitis, Allergic Contact
Keywords: Dermatitis, Allergic Contact; azithromycin; erythromycin
MeSH Terms: conditions — Dermatitis, Allergic Contact | interventions — Erythromycin; Azithromycin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- healthy individuals with erythromycin skin test: The researchers injected 30 units of erythromycin into the inner right wrist of the subjects, which is a liquid dosage form.
  Interventions: Drug: Erythromycin
- healthy individuals with azithromycin skin test: The researchers injected 30 units of azithromycin into the inner right wrist of the subjects, which is a liquid dosage form.
  Interventions: Drug: Azithromycin
- healthy individuals with physiological saline: The researchers injected 10-20 μl of physiological saline into the inner left wrist of the subjects, which is a liquid dosage form.
  Interventions: Other: physiological saline

INTERVENTIONS:
Drug: Erythromycin — The researchers injected 30 units of erythromycin into the inner right wrist of the subjects, which is a liquid dosage form.
  Groups: healthy individuals with erythromycin skin test
Drug: Azithromycin — The researchers injected 30 units of azithromycin into the inner right wrist of the subjects, which is a liquid dosage form.
  Groups: healthy individuals with azithromycin skin test
Other: physiological saline — The researchers injected 10-20 μl of physiological saline into the inner left wrist of the subjects, which is a liquid dosage form.
  Groups: healthy individuals with physiological saline

SUMMARY:
Clinical side effects of macrolides in addition to the common gastrointestinal reactions, recently it has been found that the incidence of local reactions after injection is relatively high, such as pain and itching and local inflammation. Severe skin reactions include erythema multiforme, acute systemic eruption impetigo, Stevens-Johnson syndrome, toxic epidermal necrolysis, and drug reactions with eosinophilia and systemic symptoms. The clinical study is a single-center, randomized, open, single-dose trial design. The clinical study plans to enroll 30 subjects to evaluate the incidence and severity of pain and pruritus after a single skin test in healthy subjects. A total of 30 subjects were randomly divided into 2 groups with 15 cases in each group. Erythromycin or azithromycin skin test will be performed on the left hand, and the same amount of normal saline will be injected into the right hand as the control. This clinical observation experiment helps improve the side effects and promotes upgrading macrolide antibiotics during clinical application.

ELIGIBILITY:
Inclusion Criteria:

* The age range of the subjects is from 18 to 65 years old, and there is no gender restriction for the subjects;
* Male subjects weigh more than 50kg (including 50kg) and female subjects weigh more than 45kg (including 45kg); Body mass index [BMI= weight (kg)/ height (m) 2] is in the range of 19-26 kg/m 2, including the critical value;
* The physical examination, laboratory examination, 12 lead electrocardiogram, chest X-ray (anterior lateral and lateral), and vital sign examination of the subjects are all within normal range or abnormal;
* The subjects' blood routine, blood biochemistry, and urine routine are within the normal range;

Exclusion Criteria:

* People have a clinical history of the following diseases (including but not limited to gastrointestinal, cardiovascular, musculoskeletal, endocrine, hematological, psychiatric, renal, liver, bronchial, neurological, immune, lipid metabolism disorders, or known or suspected malignant tumors);
* Patients who experience abnormal bleeding within the first 6 months of screening do not meet the criteria;
* Pregnant and lactating women; Or female urine pregnancy test positive;
* Blood routine, blood biochemistry, and urine routine examination are significantly abnormal;
* Have a history of hospitalization or surgery within 6 months before screening;
* Participate in other drug clinical studies within 3 months before screening;
* Patients with a history of prescription drug abuse and illicit drug abuse or positive urine drug screening within 6 months before screening;
* A history of alcohol abuse in the 6 months before screening, that is, drinking more than 14 units of alcohol per week (1 single drink =360 mL beer or 45 mL spirits with 40% alcohol or 150 mL wine);
* During the six months before screening, individuals who smoke more than 10 cigarettes per day or test positive for nicotine in their urine;
* Within the 3 months before screening, individuals consumed more than 1 liter of strong tea, coffee, and/or caffeinated beverages per day;
* Within 3 months before screening, the patient has a history of blood donation or acute blood loss (≥ 400mL)；
* Within 2 weeks before the screening, people use prescription drugs, over-the-counter drugs, traditional Chinese patent medicines, and simple preparations or Chinese herbal medicines;
* People have a history of allergy to any of the components of the test drug (erythromycin, azithromycin, other macrolides or ketolides);
* Any other factors deemed unsuitable for participation in this study by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study is conducted in healthy adults aged 18-65 years， and there is no gender restriction for the subjects.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Determine the occurrence of type 1 hypersensitivity reaction | 20-30 minutes after injection
  The results are observed within 20 ~ 30 minutes after antigen stimulation. The injection site of the drug is compared with normal saline. The subjects observed whether the injection site of the skin had redness, wind mass and redness, and the time of wind mass bulge and disappearance. Participants are surveyed by questionnaire for the presence and extent of pain and pruritus.
Determine the occurrence of type 4 hypersensitivity reaction | 48-72 hours after injection
  The results are observed within 48-72 hours after antigen stimulation. The injection site of the drug is compared with normal saline. The subjects observed whether the injection site of the skin had redness, wind mass and redness, and the time of wind mass bulge and disappearance. Participants are surveyed by questionnaire for the presence and extent of pain and pruritus.

CONTACTS AND LOCATIONS:
Overall Officials: Yunzhao Xu, Study Director — Affiliated Hospital of Nantong University